CLINICAL TRIAL: NCT06647797
Title: Enhancing Communication on Relationship Preservation, Safer Conception and PrEP to Promote HIV Testing in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Makerere University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Emily Hurley, Doctoral Research Faculty, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00002400; 5R34MH132473 (NIH)
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: HIV; Antenatal Care; Antiretroviral Therapy; Pre-Exposure Prophylaxis
Keywords: Antiretroviral medication

STUDY DESIGN:
Intervention Model Description: Two hospital sites. One randomized to implement the communication intervention, the other continuing with usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication intervention "HOPE" (Experimental): * Patient-facing education materials
  * Provider counseling job aid and training
  Interventions: Behavioral: HOPE Clinical Communication Campaign
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: HOPE Clinical Communication Campaign — * Patient-facing educational materials
  * Provider counseling training and job aid
  Arms: Communication intervention "HOPE"

SUMMARY:
Our novel communication strategy aims to promote HIV testing in Uganda with reassuring messages about the ability to have stable relationships and healthy families with the increased availability of pre-exposure prophylaxis (PrEP). We will evaluate the feasibility and acceptability of this communication strategy among clients and partners within assisted partner notification and antenatal care programs in two hospitals and evaluate preliminary effects.

DETAILED DESCRIPTION:
Optimizing uptake of HIV testing is critical to meeting 95-95-95 goals in sub-Saharan Africa. As 30% of new infections in occur within married or cohabitating couples, maximizing testing among individuals who are or may someday be in serious heterosexual relationships has been identified as one of the most cost-effective strategies to curb the epidemic. Childbearing is highly valued throughout Sub-Saharan Africa, and fears of relationship dissolution and loss of the ability to have children remain significant barriers to HIV testing. The expanding availability of pre-exposure prophylaxis (PrEP) presents an opportunity to counter these fears with strategic communication (NOT-MH-21-105) that reassure couples of their ability to have a healthy family even if one or both members are HIV positive. Our long-term objective is to leverage the growing availability of PrEP to determine if and how a communication strategy focused on relationship preservation and safer conception can increase testing and entry into treatment (antiretroviral therapy) or prevention (PrEP) among partnered individuals in Uganda. We recently successfully piloted this communication strategy within Uganda's assisted partner notification program (APN). In this R34, we will: (1) conduct formative research to expand the communication strategy into a multi-component intervention with broader reach; and (2) conduct a pilot trial of the intervention, PrEPing Healthy Families. To achieve Aim 1, we will work with a community advisory board (CAB) of providers to a) create communication materials (brochures, scripts) and counseling protocols tailored to clients and partners across the array of couples' testing pathways in APN and antenatal care (ANC). As CAB providers pilot materials and tracking systems with clients and partners during this development phase, study staff will conduct field observations and qualitative interviews focused on feasibility and acceptability, informing revised intervention materials. To achieve Aim 2, we will collect baseline data at APN and ANC clinics within two large public healthcare facilities over nine months. Sites will then be randomized to implement PrEPing Healthy Families or their existing communication approach (usual care) over the next nine months. We will collect mixed-methods data on feasibility and acceptability through intervention tracking in APN/ANC registers, client exit surveys, and qualitative interviews with clients, partners and providers. Through register extraction, we will examine limited efficacy on outcomes that would be relevant to a larger trial (partner HIV testing, client service uptake initiation of PrEP/ART), and explore potential moderators. Overall, results will yield important insights in a promising new communication strategy (NOT-MH-21-105) that may connect more individuals to the HIV cascades of care for treatment or prevention and prepare us for a large-scale, cluster randomized controlled trial to determine impact on testing and initiation of PrEP/ART.

ELIGIBILITY:
Inclusion Criteria:

* Client or partner of client receiving antenatal or assisted partner notification services at one of two study hospitals (Gombe Hospital or Mityana Hospital)

Exclusion Criteria:

* Individuals under the age of 18 years (for interviews and surveys only)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7666 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Change in rate of partner HIV testing (antenatal care) | 7 month baseline period and 7 month intervention period
Change in rate of partner HIV testing (assisted partner notification) | 7 month baseline period and 7 month intervention period

SECONDARY OUTCOMES:
Change overall facility-level HIV testing | 7 month baseline period and 7 month intervention period
Change in PrEP uptake among eligible HIV negative partners | 7 month baseline period and 7 month intervention period
Change in ART uptake among eligible HIV positive partners | 7 month baseline period and 7 month intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Emily Hurley, PhD, Principal Investigator — Children's Mercy Kansas City
Locations (2):
- Uganda (2):
  - Gombe Hospital, Gombe
  - Mityana Hospital, Mityana

IPD SHARING:
Plan to Share IPD: Yes
De-identified dataset and other materials will be made available to individual researchers upon reasonable request.